CLINICAL TRIAL: NCT01892215
Title: Blood Loss During Cesarean Section. Comparing Two Techniques of Blunt Expansion of Uterine Incision: Transversal vs. Cephalad-caudad. A Randomized, Controlled Trial.
Brief Title: Blood Loss During Cesarean Section. Comparing Two Techniques of Blunt Expansion of Uterine Incision: Transversal vs. Cephalad-caudad,
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of Research, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHST2012-08
Record Dates: First submitted 2013-06-30; First posted 2013-07-04 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Blunt Expansion of the Uterine Incision
Keywords: Uterine incision.; Blunt transversal expansion.; Blunt cephalad-caudad expansion.

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cephalad-caudad (Experimental): Blunt expansion of the uterine incision by the physician separating the fingers in a cephalad-caudad direction.
  Interventions: Procedure: Cephalad-caudad expansion
- Transversal expansion (Experimental): Blunt expansion of the uterine incision by the physician separating the fingers in a transversal direction.
  Interventions: Procedure: Transversal expansion

INTERVENTIONS:
Procedure: Cephalad-caudad expansion — Blunt expansion of the uterine incision by the physician separating the fingers in a cephalad-caudad direction.
  Arms: Cephalad-caudad
Procedure: Transversal expansion — Blunt expansion of the uterine incision by the physician separating the fingers in a transversal direction.
  Arms: Transversal expansion

SUMMARY:
Obstetrical blood loss is an important reason of maternal morbidity and mortality. Because of the increase in the rate of cesarean section, any procedure that could help reduce blood loss during cesarean section should be investigated. The purpose of this study was to compare 2 methods of blunt expansion of the uterine incision at the time of cesarean delivery: transversal vs. cephalad-caudad.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* Gestational age: 34 weeks or more
* Delivery by cesarean section
* Presurgical hemoglobin > 10.5 g/dL

Exclusion Criteria:

* Two or more previous cesarean sections
* History of uterine rupture in a previous pregnancy
* History of myomectomy
* History of abdominal trauma with an uterine lesion
* Blood dyscrasia
* Multiple pregnancy
* Placenta previa
* Abruptio placenta
* Stillbirth
* Sharp uterine expansion

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Blood loss (hemoglobin level) | 72 hours
  Difference in hemoglobin level between 24 hours pre-surgery and the hemoglobin level before leaving the hospital.

SECONDARY OUTCOMES:
Surgical complications | 72 hours
  Number of cases of surgical complications (hematomas, unintended extension of the uterine incision, need for transfusion) between the two techniques.
Unintented extension of uterine incision | 72 hours
  Number of cases of unintended extension of the uterine incision during surgery between the two techniques.
Hematoma formation | 72 hours
  Number of cases of hematoma formation during or after between the two techniques.
Need for transfusion | 72 hours
  Number of cases that required a blood transfusion between the two techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, MD, Principal Investigator — Saint Thomas Maternity Hospital; Alberto Morales, MD, Principal Investigator — Saint Thomas Maternity Hospital
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Panama